CLINICAL TRIAL: NCT03798704
Title: Comparison of Immunofluorescence Assay (IFA) and Chemiluminiscence Immunoassay (LIAISON®) for Diagnosis of Early Disseminated Lyme Borreliosis in Children, Younger Than 18 Years
Brief Title: Comparison of IFA and LIAISON® for Diagnosis of Early Disseminated Lyme Borreliosis in Children, Younger Than 18 Years
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Maja Arnez, izr. prof. dr. Maja Arnez, dr. med, University Medical Centre Ljubljana
Other Study IDs: Arnez 0120-134/2018
Record Dates: First submitted 2018-12-17; First posted 2019-01-10 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Lyme Disease
Keywords: Lyme disease; IFA; LIAISON; children; Slovenia
MeSH Terms: conditions — Lyme Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: IFA, LIAISON — Comparison of two diagnostic serological tests - IFA and LIAISON.

SUMMARY:
The aim of this study is to compare two different serological tests, IFA and LIAISON, for detection of Borrelia burgdorferi sensu lato IgM and IgG antibiodies in children with early disseminated Lyme borreliosis.

DETAILED DESCRIPTION:
Slovenia is highly endemic region for Lyme borreliosis (LB). LB is a tick - borne multisystem infectious disease caused by Borrelia burgdorferi sensu lato.

Solitary erythema migrans (SEM) is a typical clinical manifestation of early localized LB and microbiological confirmation of borrelial infection is not required for diagnosis.

Clinical manifestations of early disseminated LB (multiple erythema migrans (MEM), peripheral facial palsy and meningitis) are not characteristic enough to enable a reliable diagnosis, indicating the need for laboratory demonstration of borrelial infection which is mainly accomplished with serological tests.

For detection of borrelial antibodies several methods are used, such as immunofluorescent assay (IFA), enzyme immunoassay (EIA) and immunoblots. Serological tests are not standardized and have limited sensitivity and specificity.

The aim of this study is to specify and compare the sensitivity of IFA and LIAISON serological tests in early disseminated LB in children in Slovenia.

The secondary aim is to determine the influence of early antibiotic treatment of early disseminated LB on serological results in children with LB in Slovenia and to compare the serological results in children who are treated with antibiotics immediately and those who are treated later in the course of the study.

ELIGIBILITY:
Children younger than 18 years with early disseminated Lyme disease:

* multiple erythema migrans
* peripheral facial nerve palsy
* lymphocytic meningitis

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Younger then 18 years
Sampling Method: Non-Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity IFA vs. LIAISON | 2 years
  LIAISON test (E/ml) is expected to be more sensitive than IFA (titer) in detection of Borrelial antibodies in children with early disseminated LB. In all patients both asseys (LIAISON and IFA) are going to be done from the same samples. The difference in the proportion of positive tests between the two assays will be statisticaly analyzed for IgM and IgG antibodies of each patient group. P values < 0,05 will be interpreted as statistically significant.
  IFA: Titres >256 in serum and >4 in CSF will be considered positive. LIAISON values in serum: the values of IgM and IgG in serum <18 in <10 E/ml will be considered as negative, 18-22 and 10-15 E/ml will be considerd as border values and >22 in >15 E/ml will be considered as positive.
  LIAISON in cerebral fluid: the values of IgM in IgG in cerebral fluid <2,5 and <4,5 E/ml will be considered as negative, values 2,5-3,5 and 4,5-5,5 E/ml will be considered as border values and >2,5 in >5,5 E/ml will be considered as positive.

CONTACTS AND LOCATIONS:
Locations (1):
- University clinical center, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided